CLINICAL TRIAL: NCT02363322
Title: A Multicenter Randomized Safety and Efficacy Study of Putative Investigational Therapeutics in the Treatment of Patients With Known Ebola Infection
Brief Title: Putative Investigational Therapeutics in the Treatment of Patients With Known Ebola Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: The Ministry of Health and Social Welfare, Liberia (Unknown); Ministry of Health and Sanitation, Sierra Leone (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); The Ministry of Health and Public Hygiene, Guinea (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150083; 15-I-0083 (Other: NIH Office of Protocol Services)
Record Dates: First submitted 2015-02-13; First posted 2015-02-16 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-06

CONDITIONS: Ebola Virus Infection
Keywords: Medical Countermeasures; VHF; EVD
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — ZMapp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A/Current Standard of Care Alone (Active Comparator): A/Current Standard of Care Alone: Optimized standard of care to include aggressive fluid resuscitation, hemodynamic support, and other interventions available in an optimized care setting
  Interventions: Other: A/Current Standard of Care Alone
- B/Current Standard of Care Plus ZMapp (Experimental): B/Current Standard of Care Plus ZMapp: ZMapp (Trademark) + Optimized standard of care to include aggressive fluid resuscitation, hemodynamic support, and other interventions available in an optimized care setting.
  ZMapp 50mg/kg IV administered every third day for 3 infusions.
  Interventions: Drug: B/Current Standard of Care Plus ZMapp; Other: A/Current Standard of Care Alone

INTERVENTIONS:
Drug: B/Current Standard of Care Plus ZMapp — Triple monoclonal cocktail of antibodies against Zaire species of Ebola virus
  Arms: B/Current Standard of Care Plus ZMapp
Other: A/Current Standard of Care Alone — Optimized standard of care for Ebola virus infection

SUMMARY:
Background:

- Ebola is a viral infection that can spread quickly and causes life-threatening disease. Right now there is an Ebola outbreak in many countries in West Africa. There are no approved treatments for Ebola. But possible treatments are being developed. Researchers need to study these treatments to see if they help people get better.

Objective:

- To identify possible Ebola treatments. Also, to learn if adding 1 or more experimental drugs to advanced Ebola care can reduce the risk of death.

Eligibility:

- People who have recently been diagnosed with Ebola, usually by a test called the Polymerase Chain Reaction (PCR), and have been hospitalized in an isolation unit for treatment.

Design:

* Participants will be randomly assigned to Group A or B. Both groups will get advanced level care. One group will also get an experimental drug.
* Participants may have blood tests. They may have another PCR test.
* Researchers will try to learn how the participant got Ebola.
* Participants put in the experimental drug group may start taking medicine within 24 hours of enrollment. It may be given by mouth or intravenously. Additional doses may be needed.
* Participants may have a series of timed blood tests over the first 24 to 48 hours after they take the medicine.
* Blood will be drawn frequently. Other body fluids (urine, stool, vaginal fluid, etc.) may also be collected.
* Participants will be followed for up to 60 days. They may be evaluated for any long-term effects of the experimental treatment(s). They may be asked to return for 1 or more outpatient visits.
* For consenting participants, follow-up will be extended for up to one full year past Day 58 with contact/visits every 1-3 months to assess for a history of signs or symptoms potentially consistent with late onset of virologic relapse syndrome.

DETAILED DESCRIPTION:
Ebolaviruses (EBOV) are members of the Filoviridae and are known primarily as the underlying cause of severe viral hemorrhagic fevers with disturbingly high case fatality rates. Between 1994 and the present, there have been many EBOV outbreaks affecting mostly central Africa, with 2 large outbreaks in 1995 in Kikwit, Democratic Republic of Congo (DRC), and in Gulu, Uganda in 2000-2001. However, the 2014 West African outbreak significantly exceeds all previous outbreaks in geographic range, number of patients affected, and in disruption of typical activities of civil society.

There is strong consensus that the most important element necessary to improve survival from Ebola infection is the provision of full hemodynamic support in the form of aggressive fluid replacement, ability to diagnose and correct severe metabolic derangements, and other standards of modern medical care available in resource-rich environments. However, against this background, a small series of investigational agents or interventions have also been proposed as putative antiviral strategies of potential utility in treating this infection. Unfortunately, phase 1/2 data supporting the safety and efficacy of these agents is generally lacking, and thus there should be equipoise as to which, if any, of these interventions should be utilized in the treatment of severe infection.

In this multicenter randomized trial, we propose a flexible trial design with frequent interim monitoring to facilitate early elimination of poorly performing treatments as well as the introduction of new candidate therapies. The trial allows for a series of pairwise comparisons of novel interventions against a background of optimized medical care, with the goal of determining whether one or more of these interventions can improve the mortality over that achievable through optimized standard-of- care (oSOC) alone. The primary endpoint of this trial will be comparative mortality at Day 28, with a number of secondary endpoints that hopefully will generate generalizable knowledge about the relative safety and antiviral activity of these adjunctive interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males or females with documented positive PCR for Ebola virus infection within 10 days of enrollment
* Willingness of study participant to accept randomization to any assigned treatment arm
* Access to oSOC
* All males and females of childbearing potential, must be willing to use highly effective methods of contraception [e.g. absolute abstinence from potentially reproductive sexual activity, hormonal, surgical or multiple barrier/combined], from time of enrollment for the duration of study participation.
* Must agree not to enroll in another study of an investigational agent prior to completion of last required protocol visit (Day 58)
* Ability to provide informed consent personally, or by a legally-authorized [per applicable local laws and regulations] representative [LAR] if the patient is unable to do so.

EXCLUSION CRITERIA:

* Any medical condition that, in the opinion of the site investigator, would place the patient at an unreasonably increased risk through participation in this study, including any past or concurrent conditions that would preclude randomization to one or more of the assigned treatment arms.
* Prior treatment with any investigational antiviral drug therapy against Ebola infection other than experimental vaccines, within 5 half-lives or 30 days, whichever is longer, prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (11):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- CTE Forecariah, Forécariah, Guinea
- Liberia (2):
  - Monrovia Medical Unit, Monrovia
  - ELWA III Hospital, Paynesville
- Sierra Leone (7):
  - Police Training School 1 (PTS1), Western Rural District, Freetown
  - Emergency Ebola Treatment Unit, Goderich
  - Police Training School 2, Hastings
  - Chinese Friendship Hospital, Jui
  - International Medical Corps (IMC) Kambia, Kambia
  - International Medical Corps (IMC) Lunsar, Port Loko
  - Adventist Development and Relief Ebola Treatment Unit, Waterloo

REFERENCES:
- [Background] Joffe S. Evaluating novel therapies during the Ebola epidemic. JAMA. 2014 Oct 1;312(13):1299-300. doi: 10.1001/jama.2014.12867. No abstract available. PMID 25211645
- [Background] Kanapathipillai R. Ebola virus disease--current knowledge. N Engl J Med. 2014 Sep 25;371(13):e18. doi: 10.1056/NEJMp1410741. No abstract available. PMID 25251632
- [Background] Piot P, Muyembe JJ, Edmunds WJ. Ebola in west Africa: from disease outbreak to humanitarian crisis. Lancet Infect Dis. 2014 Nov;14(11):1034-1035. doi: 10.1016/S1473-3099(14)70956-9. Epub 2014 Oct 1. No abstract available. PMID 25282665
- [Derived] PREVAIL II Writing Group; Multi-National PREVAIL II Study Team; Davey RT Jr, Dodd L, Proschan MA, Neaton J, Neuhaus Nordwall J, Koopmeiners JS, Beigel J, Tierney J, Lane HC, Fauci AS, Massaquoi MBF, Sahr F, Malvy D. A Randomized, Controlled Trial of ZMapp for Ebola Virus Infection. N Engl J Med. 2016 Oct 13;375(15):1448-1456. doi: 10.1056/NEJMoa1604330. PMID 27732819
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0083.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginnning in March 2015 through November 2015 a total of 72 patients were enrolled at sites in Liberia, Sierra Leone, Guinea, and the United States.
Groups:
- A/Current Standard of Care Alone: Optimized standard of care to include aggressive fluid resuscitation, hemodynamic support, and other interventions available in an optimized care setting
  Treatment A: Optimized standard of care for Ebola virus infection
- B/Current Standard of Care Plus ZMapp: ZMapp (Trademark) + Optimized standard of care to include aggressive fluid resuscitation, hemodynamic support, and other interventions available in an optimized care setting.
  ZMApp: Triple monoclonal cocktail of antibodies against Zaire species of Ebola virus
Period: Overall Study
Arm/Group | A/Current Standard of Care Alone | B/Current Standard of Care Plus ZMapp
Started | 36 | 36
Completed | 35 | 36
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- A/Current Standard of Care Alone: Optimized standard of care to include aggressive fluid resuscitation, hemodynamic support, and other interventions available in an optimized care setting
- Total: Total of all reporting groups
Arm/Group | A/Current Standard of Care Alone | B/Current Standard of Care Plus ZMapp | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (16.4) | 24.3 (18.3) | 26.1 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 40
  Male | 19 | 13 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 29 | 60
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  Liberia | 2 | 3 | 5
  United States | 1 | 0 | 1
  Guinea | 5 | 7 | 12
  Sierra Leone | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Death at Day 28
Time Frame: 28 days
Population: Seven of the eight deaths recorded in ZMapp recipients occurred before day 4, before the second of three planned infusions of ZMapp. The exception was one patient who received a second infusion on day 4 and died later that day. In the group that received the current standard of care alone, all 13 deaths occurred during the first 8 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | A/Current Standard of Care Alone | B/Current Standard of Care Plus ZMapp
Number analyzed (Participants) | 35 | 36
Participants | 13 | 8

2. Secondary Outcome: Number of Participants With ZMapp Infusion-related Adverse Events
Description: Adverse events related to ZMapp infusions
Time Frame: 10 Days
Population: Arm A Received the Current Standard of Care Alone and not the ZMapp infusion
Measure: Number; unit: participants
Arm/Group | A/Current Standard of Care Alone | B/Current Standard of Care Plus ZMapp
Number analyzed (Participants) | 0 | 36
participants
  Hypotension |  | 7
  Elevation in fever |  | 8
  Tachycardia |  | 4
  Tachypnea |  | 3
  Hypertension |  | 3
  Confusion |  | 2
  Seizure |  | 1
  Difficulty Breathing |  | 1
  Chills |  | 1
  Vomiting |  | 1
  Agitation |  | 1

3. Secondary Outcome: Plasma Viral Load
Description: Time to viral clearance
Time Frame: 28 days
Measure: Median (Full Range); unit: days
Arm/Group | A/Current Standard of Care Alone | B/Current Standard of Care Plus ZMapp
Number analyzed (Participants) | 35 | 36
days | 13 [0 to 28] | 9 [0 to 28]

ADVERSE EVENTS:
Time Frame: 8 months, from March 2015 through November 2015
Description: Only Serious Adverse Events and Infusion related events were recorded.
Arm/Group | A/Current Standard of Care Alone | B/Current Standard of Care Plus ZMapp
All-Cause Mortality (participants affected / at risk) | 13/35 | 8/36
Serious Adverse Events (participants affected / at risk) | 13/35 | 11/36
Other Adverse Events (participants affected / at risk) | 0/35 | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/Current Standard of Care Alone (N=35) | B/Current Standard of Care Plus ZMapp (N=36)
Worsened renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Death due to Hypotensive Shock (Vascular disorders) | 1 (1) | 0 (0)
Death due to EVD (Infections and infestations) | 10 (10) | 2 (2)
Head Injury (Nervous system disorders) | 1 (1) | 0 (0)
Multi-organ failure due to EVD (Infections and infestations) | 2 (2) | 3 (3)
Death due to sepsis (Infections and infestations) | 0 (0) | 1 (1)
Generalized seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypovolemic shock due to acute hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Severe diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arterial Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hospitalization with febrile illness (malaria) (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/Current Standard of Care Alone (N=35) | B/Current Standard of Care Plus ZMapp (N=36)
Hypotension (Vascular disorders) | NA | 7 (7)
Elevation in Fever (Infections and infestations) | NA | 8 (8)
Tachycardia (Vascular disorders) | NA | 4 (4)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | NA | 3 (3)
Hypertension (Vascular disorders) | NA | 3 (3)
Confusion (Nervous system disorders) | NA | 2 (2)
Seizure (Nervous system disorders) | NA | 1 (1)
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Chills (Infections and infestations) | NA | 1 (1)
Vomiting (Gastrointestinal disorders) | NA | 1 (1)
Agitation (Nervous system disorders) | NA | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the severity of the underlying illness (Ebola infection) only infusion-related adverse events were captured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT02363322/Prot_SAP_ICF_000.pdf